CLINICAL TRIAL: NCT03660046
Title: A Prospective Cohort Study Evaluating the Impact of Three Progestin-based Hormonal Contraceptive (HC) Methods on Immunologic Changes in the Female Genital Tract (FGT) and Systemically
Brief Title: Contraceptive Hormones, Immunity, and Microbiome Evaluation
Acronym: CHIME
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alicia K Smith, Associate Professor, Emory University
Other Study IDs: IRB00104017; R01HD095741-01A1 (NIH)
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hormonal Contraception
Keywords: Human immunodeficiency virus; Sexually Transmitted Diseases; Contraceptives
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Medroxyprogesterone Acetate; etonogestrel; Levonorgestrel; Copper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Depot medroxyprogesterone acetate (DMPA): This arm includes subjects that choose Depot medroxyprogesterone acetate (DMPA) as contraception.
  Interventions: Drug: Depot medroxyprogesterone acetate (DMPA)
- Etonogestrel implant (Eng-Implant): This arm includes subjects that choose Etonogestrel implant (Eng-Implant) as contraception.
  Interventions: Drug: Etonogestrel implant (Eng-Implant)
- Levonorgestrel IUD (Lng-IUD): This arm includes subjects that choose Levonorgestrel Intrauterine device (Lng-IUD) as contraception.
  Interventions: Drug: Levonorgestrel IUD (Lng-IUD)

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate (DMPA) — Depot medroxyprogesterone acetate (DMPA) will be dispensed from the Grady Pharmacy Service and will be administered every 12 weeks at the standard dose of 150 mg Intramuscular injection, beginning from week 3 of study enrollment and repeated every 13 weeks
  Other Names: Medroxyprogesterone acetate (MPA); Depo-Provera
  Groups: Depot medroxyprogesterone acetate (DMPA)
Drug: Etonogestrel implant (Eng-Implant) — A standard Nexplanon rod Implant that is a subdermal implant in the arm. This will be placed at study week 3 by Dr. Haddad or a trained clinician. It contains Etonogestrel 68mg.
  Other Names: Nexplanon
  Groups: Etonogestrel implant (Eng-Implant)
Drug: Levonorgestrel IUD (Lng-IUD) — The Levonorgestrel Intrauterine Device (Lng-IUD) (Mirena or copper) will be placed at study week 3 by Dr. Haddad or a trained clinician.
  Other Names: Mirena; Copper
  Groups: Levonorgestrel IUD (Lng-IUD)

SUMMARY:
The study is a prospective cohort study to explore the mechanisms underlying the HIV risk associated with pharmacologic doses of exogenous sex hormones via hormonal contraceptives specially progestin-containing hormonal contraception (HC). The study seeks to test that HC induce immunologic changes capable of altering HIV susceptibilities, that these effects will vary by contraceptive type, and that they will be modified by the vaginal microenvironment.

DETAILED DESCRIPTION:
This study is a translational research project to explore the mechanisms underlying the HIV risk associated with pharmacologic doses of exogenous sex hormones (via hormonal contraceptives). Emerging data suggests that certain hormonal contraceptives may induce mucosal and systemic immune changes that could increase the risk of infection with HIV. While several studies have aimed to characterize immunologic changes in women using hormonal contraceptives, the nature and the magnitude of these immune changes have not been adequately defined due to limitations in study design rigor, and small and statistically underpowered sample sizes.

The study will prospectively recruit cohorts of HIV-uninfected women initiating hormonal contraception to characterize systemic and lower genital tract innate and adaptive immunologic changes that occur over a course of up to 4 months. This study will test the overarching hypothesis that hormonal contraceptives induce systemic and mucosal immune changes capable of altering susceptibilities and/or responses to diseases including HIV infection, and that these effects vary markedly in nature and magnitude by contraceptive type and will be modified by the vaginal microenvironment. The main aim is to determine the immunologic alterations in female genital and systemic immune profile associated with depot medroxyprogesterone acetate (DMPA), Etonogestrel implant (Eng-Implant) and Levonorgestrel IUD (Lng-IUD).

ELIGIBILITY:
Inclusion Criteria:

* Female sex, defined by sex at birth.
* Age ≤ 45 years. If < 18 years of age, participant must be capable of providing assent, understanding and complying with all study procedures, and have written informed consent from a parent or legal guardian.
* Normal menses (occurring within 22-35 day intervals) for > 2 cycles. Women who are postpartum or post-abortion who have resumed menses are eligible.
* Intact uterus and cervix.
* Interested in initiating HC and willing to accept DMPA, Eng-Implant or Lng-IUD.
* Willing to delay initiation of HC for up to 1 month.
* Able and willing to provide informed consent, and undergo study procedures.
* Negative HIV test by Ora-Quick© method at Screening Visit.
* Agree to abstain from vaginal intercourse or using intra-vaginal products for 1 day prior to each study visit.

Exclusion Criteria:

* Pregnant or planning to become pregnant within the next year.
* Breastfeeding, if not having active menstrual cycles. Breastfeeding is not exclusionary if the participant is actively cycling.
* History of loop electrosurgical excision procedure (LEEP), conization, or cryosurgery within the past year.
* Current use of systemic HC or IUD, based on self-report and/or hormonal testing.
* Taking concurrent medications that interact with selected HC.
* Contraindications to selected contraceptive per the Center for Disease Control medical eligibility criteria or judgment of clinician.
* Allergy to lidocaine for cervical biopsies (if consenting to optional biopsies).

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female sex, defined by sex at birth
Study Population: Participants will be selected from several sites in the greater Atlanta community to include: family planning clinics, OB/GYN practice/reproductive heath clinics, community based recruitment through postings at community centers, community health fairs, coffee shops and local universities, as well as web-based recruitment through the national ResearchMatch.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Change in mean total leukocytes and CD4+ T-cells expressing CCR5 in the lower female genital tract (FGT) among the three intervention groups pre and post contraception | Week 1 and Week 3 (pre contraception), and 13 and 15 weeks after initiating contraception
  Using Fortessa flow cytometer and Luminex, effector memory Cluster Differentiation 4 (CD4) + Thymocytes (T) cells will be analyzed for surface expression of HIV coreceptors cell surface receptor C-C chemokine receptor type 5 (CCR5) and reported as percent of total leukocytes and CD4+ T-cells. The cytometry will use the cervicovaginal fluid (CVF) collected by cervicovaginal lavage (CVL).This test will characterize the alterations in female genital and systemic immune profiles associated with three long-acting progestin-only Hormonal Contraception.
Change in Nugent's score among the three intervention groups pre and post contraception | Week 1 and Week 3 (pre contraception), and 13 and 15 weeks after initiating contraception
  The Nugent Score is a Gram stain scoring system for vaginal swabs to diagnose bacterial vaginosis. The Nugent score is calculated by assessing for the presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0 to 4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0 to 4), and curved Gram-variable rods (Mobiluncus spp. morphotypes; scored as 0 to 2). A score of 7 to 10 is consistent with bacterial vaginosis without culture.
Percent of expression of 16S rRNA gene sequencing among the three intervention groups pre and post contraception | Week 1 and Week 3 (pre contraception), and 13 and 15 weeks after initiating contraception
  16 Svedberg ribosomal RNA (16S rRNA) is the component of the 30 Svedberg ribosomal RNA (30S rRNA) small subunit of a prokaryotic ribosome that binds to the Shine-Dalgarno sequence. The genes coding for it are referred to as 16S rRNA gene and are used in reconstructing phylogenies. 16S rRNA gene sequence analysis can better identify poorly described, rarely isolated, or phenotypically aberrant strains, can be routinely used for identification of mycobacteria, and can lead to the recognition of novel pathogens and uncultured bacteria.The term 16S refers to how it settles to when centrifuged (it's called a sedimentation rate, and it's measured in Svedberg (S) units).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Smith, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Health System, Atlanta, Georgia
  - The Emory Clinic, Bldg A., 2nd Floor, 1365 Clifton Road, NE, Atlanta, Georgia
  - Atlanta Women's Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No